CLINICAL TRIAL: NCT06850545
Title: Kuopio Lutetium-177 Study in Patients with PSMA-Positive Metastatic Prostate Cancer
Acronym: KuPSMALu
Status: Recruiting | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Okko Kääriäinen, Clinical oncologist, Kuopio University Hospital
Other Study IDs: KUH5654217
Record Dates: First submitted 2025-02-22; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Prostate Adenocarcinoma; PSMA PET-Positive Castration-Resistant Prostate Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — cfDNA samples during the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
KuPSMALu-trial is an observational study for patients treated with 177LuPSMA-I&T in Kuopio University Hospital, Finland. Study focuses on efficacy, safety and biomarker research.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must sign informed consent to participate in the study.
2. Patients must be over 18 years of age.
3. Patients must have histologically confirmed metastatic prostate adenocarcinoma. Histological samples may show neuroendocrine features, but the primary component must be adenocarcinoma.
4. Patients must have metastatic castration-resistant prostate cancer (mCRPC) that has been treated with at least docetaxel and abiraterone or enzalutamide, or the patients must have declined chemotherapy or be ineligible for docetaxel-based chemotherapy due to contraindications.
5. Patients must have an adequate performance status: WHO 0-2.
6. Castration must have been achieved either chemically (LHRH analog or antagonist) or surgically (orchiectomy). Castration is defined as a low testosterone level (S-testosterone ≤ 1.7 mmol/l).
7. Patients must have PSMA-positive tumor burden detected by 18F-PSMA-PET-CT imaging.
8. Patients must have adequate renal and liver function (Creatinine < 2x upper limit of normal (ULN), ALT and ALP < 5x ULN).
9. Patients' blood counts must be within acceptable levels (Hb ≥ 100 g/l, Platelets ≥ 100 x 10⁹/L, Leukocytes ≥ 3.0 x 10⁹/L, or Neutrophils ≥ 1.0 x 10⁹/L).
10. The expected survival must be more than 6 months.
11. Patients with ejaculatory capacity must commit to not donating sperm during the treatments and for 6 months after treatment completion.

Exclusion Criteria:

1. Patients whose physical condition and cooperation are insufficient to follow the given instructions.
2. Patients who do not meet the criteria mentioned in the inclusion criteria.
3. Patients must not have PSMA-negative tumor burden in the liver. The amount of PSMA-negative tumor burden must not exceed the amount of PSMA-positive tumor burden.
4. Patients with symptomatic untreated spinal cord compression.
5. Patients must not have acute hydronephrosis or urinary tract obstruction.
6. Patients must not have a recurrent infection that impairs functional capacity.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mCPRC patients treated with 177LuPSMA-I&T in Kuopio University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Overall survival in the trial

SECONDARY OUTCOMES:
PSA decrease of 50% or more | 36 weeks
  PSA decrease of 50% or more within the treatment period
Adverse Events | 36 weeks
  Treatment-related grade ≥3 and serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: No